CLINICAL TRIAL: NCT06928012
Title: Risk Factors , Types and Neuroimaging Findings in Patients With Cerebral Palsy at Assiut University Children's Hospital
Acronym: cerebral palsy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Naser Abd El Fadeel Ali, Principal investigator, Assiut University
Other Study IDs: Cerebral palsy neuroimaging
Record Dates: First submitted 2025-03-22; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Cerebral palsy (CP) is the most common motor disorder among children as its worldwide prevalence is ranging from 1.5 to more than 4 per 1000 live births or children of a defined age range.

* Pediatric cerebral palsy is a clinical syndrome caused by brain injury or lesions in children from before birth to 1 month after birth, and mainly manifests as non progressive central dyskinesia and abnormal posture.
* Research has shown that the prevalence of cerebral palsy in children worldwide is about 3.16% , and results in heavy familial and social burdens as well as usage of medical resources, Despite considerable research , the complex etiology and pathogenesis of cerebral palsy remain unclear. The high-risk factors of cerebral palsy are complex and diverse (CP) appeared to be more prevalent in low- or middle-income countries than in high-income countries.

(CP) prevalence was about 3.6 and 2.9 per 1000 children in Uganda and Egypt, respectively, but the prevalence was 1.8 to 2.3 cases per 1000 children in the USA, Europe, and Australia.

-Cerebral palsy (CP) describes a group of disorders of the development of movement and posture, causing activity limitation, that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain. It begins in early childhood and persists through the lifespan.

It was first reported as a movement disorder in the historical documents of the Sumerians, and Hippocrates.

-Cerebral palsy (CP) is the major cause of motor impairment in young children, The clinical picture changes over time, and a recent review showed that referral for diagnosis typically happens between 10 and 21 months of age.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common motor disorder among children as its worldwide prevalence is ranging from 1.5 to more than 4 per 1000 live births or children of a defined age range.

* Pediatric cerebral palsy is a clinical syndrome caused by brain injury or lesions in children from before birth to 1 month after birth, and mainly manifests as non progressive central dyskinesia and abnormal posture.
* Research has shown that the prevalence of cerebral palsy in children worldwide is about 3.16% , and results in heavy familial and social burdens as well as usage of medical resources, Despite considerable research , the complex etiology and pathogenesis of cerebral palsy remain unclear. The high-risk factors of cerebral palsy are complex and diverse (CP) appeared to be more prevalent in low- or middle-income countries than in high-income countries.

(CP) prevalence was about 3.6 and 2.9 per 1000 children in Uganda and Egypt, respectively, but the prevalence was 1.8 to 2.3 cases per 1000 children in the USA, Europe, and Australia.

-Cerebral palsy (CP) describes a group of disorders of the development of movement and posture, causing activity limitation, that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain. It begins in early childhood and persists through the lifespan.

It was first reported as a movement disorder in the historical documents of the Sumerians, and Hippocrates.

-Cerebral palsy (CP) is the major cause of motor impairment in young children, The clinical picture changes over time, and a recent review showed that referral for diagnosis typically happens between 10 and 21 months of age.

Even patients with the same motor impairment are not the same, and that is why the development of functional scales has been an important step in management of (CP) patients .

children with cerebral palsy, is developed to measure change in gross motor function over time. Both the GMFCS feature a 5-level ordinal scale which reflects, in a decreasing order, the level of independence and functionality of children with CP.

-Etiology and Pathogenesis of cerebral palsy remain unclear. The high-risk factors of cerebral palsy are complex and diverse and the time span of these risk factors is long, which can occur at birth as well as before or after birth. Moreover, these risk factors affect each other and form an intertwined network, leading to the occurrence of diseases.

Many risk factors are identified during antenatal, natal, and post-natal periods, including multiple births, intrauterine infection, preterm, perinatal stroke, birth asphyxia, perinatal infection, placental pathology, and congenital malformations .

At the present time, it is unrealistic to determine and clear-categorize the cause; however, Investigators should do every possible effort to evaluate causal pathways or causes.

If there is a clear evidence indicating that a major component of the cause, or the cause was operative in a certain time window, so insult timing could be determined, as a previously well infant with post-natal meningitis. However, it is important to record adverse events during pregnancy and the perinatal period of cerebral palsy, and it is not sufficient to depend on the presence of such events as causes for the cerebral palsy genesis in the affected patient, Although diagnosis of cerebral palsy is mainly clinical, the American Academy of Neurology recommends all cases of cerebral palsy should undergo neuroimaging at least once, preferably MRI because of better detection rates. Neuroimaging plays a key role in clarifying etiology, determining the nature and timing of brain lesion, establishing prognosis, for the assessment of recurrence risk and genetic counseling of families and to limit unnecessary investigations

, these risk factors affect each other and form an intertwined network, leading to the occurrence of diseases Unfortunately, previous research on risk factors for cerebral palsy in children has been limited and inconsistent .

. Unfortunately, previous research on risk factors for cerebral palsy in children has been limited and inconsistent. For example, a study was limited to at-birth and fetal factors ,Perinatal factors and maternal factors are usually ignored ,Whether gestational hypertension increases the risk of cerebral palsy in children has long been controversial.

A study has pointed out that preterm birth leads to a significant increase in the incidence of cerebral palsy.

One study has also pointed to neurodevelopmental impairment, rather than preterm birth, as a risk factor for cerebral palsy .

Emergency cesarean section and premature rupture of membranes are risk factors for cerebral palsy in term infants, but the relationship between the three is not close in preterm infants. In addition, due to the development of maternal and neonatal medical and nursing techniques, the risk factors for pediatric cerebral palsy have changed, such as premature birth and the incidence of brain injury caused by hyperbilirubinemia has dropped sharply.

In today's medical context, identifying or updating risk factors for pediatric cerebral palsy can inform preventive interventions.

Aiming at the above-mentioned controversy, this study conducted a meta-analysis of the literature published over the past 20 years exploring the pregnancy risk factors of mothers with infantile cerebral palsy, in order to find the main risk factors of infantile cerebral palsy .

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy is defined as a group of permanent disorder of posture and movement resulting from a non-progressive disturbance which occurred in fetal or infant brain .
* Children ages 6 months to 16 years.

Exclusion Criteria:

* Children with identified chromosomal abnormalities or syndromatic features
* Progressive condition is identified to cause the movement, development, and posture disorder.

Ages: 6 Months to 16 Years | Sex: All
Age Groups: Child
Study Population: Cerebral patient admitted to Assiut university within one year
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of risk factors of pediatric cerebral palsy | Baseline
  to evaluate different risk factors of pediatric cerebral palsy
Evaluation of types of pediatric cerebral palsy | Baseline
  to evaluate different types of pediatric cerebral palsy
Evaluation of neuroimaging of of pediatric cerebral palsy | Baseline
  Evaluation of neuroimaging of of pediatric cerebral palsy